CLINICAL TRIAL: NCT04185376
Title: Prevalence and Risk Factors for Pelvic Floor Disorders During Pregnancy in a Cohort of Egyptian Women
Brief Title: Prevalence and Risk Factors for Pelvic Floor Disorders
Status: Completed | Type: Observational
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Sahar MY Elbaradie, associate Professor, Fayoum University Hospital
Other Study IDs: fayoum
Record Dates: First submitted 2019-11-30; First posted 2019-12-04 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A 200 patients: patients with one or more PFDs significant psychological strain in at least one pelvic floor domain
  Interventions: Other: Questionnaire
- group B 200 patients: patients without any pelvic floor complaints
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — a self-administered questionnaire for the assessment of pelvic floor disorders, their risk factors and their impact of quality of life during pregnancy and postpartum period which integrates bladder, bowel and sexual function, pelvic organ prolapse, severity, bothersomeness and conditions specific quality of life in women with urinary incontinence (UI) and/or POP. The questionnaire is divided into four main domains (bladder, bowel, pelvic organ prolapse, sexual function) and each question is scored from zero to three. The additive scores are divided by the maximum reachable score and multiplied by ten, giving a value between zero (0 = no symptoms) and ten (10 = maximum symptoms) for each of the domains.

SUMMARY:
Pelvic floor disorders (PFD) can adversely affect the quality of life of a woman and they can occur during different stages of female life such as during pregnancy, early postpartum period or during menopause. It is well known that pregnancy and vaginal birth are significant risk factors in the etiology of PFD and predicting models like UR-CHOICE score were developed for this reason to provide mothers-to-be with sufficient information regarding their subsequent risk of PFD. Pregnancy, childbirth and the immediate postpartum period, where the demands on the pelvic floor and the incidence of pelvic floor trauma are particularly high, offers an optimal opportunity for such counseling and prevention.

DETAILED DESCRIPTION:
Pelvic floor disorders (PFDs) can adversely affect the quality of life (QoL) of a woman and they can occur during different stages of female life such as during pregnancy, early postpartum period or during menopause. The reported prevalence of PFDs varies widely both during and after pregnancy and reported up to 30-50%. Besides, the term PFD includes a broad spectrum of conditions such as urinary incontinence (UI), pelvic organ prolapse (POP) or anal incontinence (AI). Many risk factors seem to be involved like the pregnancy itself, mode of delivery, parity, the use of episiotomy, obesity, increased age and so on. It is well known that pregnancy and vaginal birth are significant risk factors in the etiology of PFDs and predicting models like UR-CHOICE score were developed for this reason to provide mothers-to-be with sufficient information regarding their subsequent risk of PFD. The identification of women during their pregnancy who are at higher risk for PFD remains a key element in targeting of prevention and planning health of resource allocation strategies. Pregnancy, childbirth and the immediate postpartum period, where the demands on the pelvic floor and the incidence of pelvic floor trauma are particularly high, offers an optimal opportunity for such counseling and prevention. The validated German pelvic floor questionnaire modified for pregnancy and postpartum period is thus an important tool identifying such symptoms and helping clinicians assess patient's quality of life. The aim of the present study was to evaluate the prevalence of PFDs in a cohort of Egyptian women during pregnancy. Furthermore, we searched for clinical risk factors that correlate with the occurrence of PFDs during pregnancy in the investigator's population.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* any trimester of pregnancy
* planned delivery at our institution.

Exclusion Criteria:

* Women with the inability to complete the questionnaire

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Women ran through the questionnaire either during their first or last visit at the outpatient clinic and afterwards they were classified into two groups: patients with one or more PFDs (n = 96/200) (= significant psychological strain in at least one pelvic floor domain) and patients without any pelvic floor complaints (n = 104/200). Clinical information, including obstetrical and neonatal data
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
subjective pelvic floor-related quality of life symptoms. | one year
  the prevalence of pelvic floor disorders during pregnancy and the clinical risk factors which correlate with pelvic floor symptoms during pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- sahar M.Y elbaradie, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided